CLINICAL TRIAL: NCT00740753
Title: A Humanitarian Device Exemption Use Protocol of TheraSphere for Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: Radiolabeled Glass Beads Used for Treating Patients With Primary Liver Cancer When Surgery is Not an Option
Acronym: Y-90HDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Kenneth J Kolbeck MD PhD, Associate Professor, Charles T. Dotter Department of Interventional Radiology, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00002377; HDE 2377 (Other: Oregon Health & Science University)
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Liver Cancer; Hepatoma
Keywords: liver tumor; cancer; hepatoma; yttrium
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Other): yttrium 90 (TheraSphere) administration
  Interventions: Device: Yttrium 90 (TheraSphere)

INTERVENTIONS:
Device: Yttrium 90 (TheraSphere) — Y-90 embedded glass microspheres
  Other Names: Yttrium - 90; Y-90; TheraSphere

SUMMARY:
Fewer than 15% of hepatoma patients are suitable candidates for surgical removal of their cancer. The purpose of this protocol is to provide supervised access at Oregon Health and Science University to Y-90 treatment to provide these patients access to an alternate therapy. The radioactive beads are placed directly near or into the liver tumor with the intention of destroying the tumor cells.

DETAILED DESCRIPTION:
Patients receive Y-90 (yttrium) glass microspheres via percutaneous hepatic arterial infusion. Patients amy be retreated between 30-90 days after initial infusion. After completion of therapy, patients are followed for 30 days and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HCC
* Cancer is unresectable
* ECOG Score 0-2
* Age of 18 yrs or over
* Able to give consent

Exclusion Criteria:

* Contraindication to angiography and selective visceral catheterization
* Portal hypertension with portal venous shunt away from the liver
* Evidence of potential delivery of > 16.5 mCi of radiation to the lungs
* Evidence of any detectable Tc-99m MAA flow to the stomach or duodenum, after application of established angiographic techniques to stop such flow
* Significant extrahepatic disease representing an imminent life-threatening outcome
* Severe liver dysfunction or pulmonary insufficiency
* Active uncontrolled infection
* Significant underlying medical or psychiatric illness
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2004-08; Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Tumor response after treatment based on tumor marker and lab results, CT scan and patient's symptoms. | 2 weeks, 1 month and then every 3 months
  Tumors will decrease in size

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Kolbeck, MD, PhD, Principal Investigator — OHSU Knight Cancer Institute